CLINICAL TRIAL: NCT00194870
Title: Electroencephalography (EEG) and Deep Brain Stimulation (DBS) in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0309006367
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy
Keywords: EEG; DBS
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digital EEG (Other): Digital EEG
  Interventions: Procedure: EEG

INTERVENTIONS:
Procedure: EEG — computer-assisted analysis of the digitally-recorded EEG signals

SUMMARY:
Patients with epilepsy undergoing deep brain stimulation (DBS) have electroencephalograms (EEGs) recorded before and during their stimulation treatment. Subsequently the investigators will be using computer-assisted analysis of the digitally-recorded EEG signals to assess the effects of DBS on the brain-wave frequency content and any abnormal seizure-like patterns that may be present.

DETAILED DESCRIPTION:
Study Purpose:

The purpose of this study is to assess EEG changes during electrical stimulation of the thalamus to treat people with epilepsy.

Background on stimulation of the anterior nucleus of the thalamus for epilepsy:

Of the estimated 4 million people in the U.S. and Europe with epilepsy, approximately 1.2 million have recurrent seizures that do not respond to antiepileptic drugs. For these patients, alternative treatments consist of neurosurgical removal of the seizure source from the brain, or surgical implantation of a device to electrically stimulate the vagus nerve in the neck. In spite of these options, a significant number of people suffer from seizures that remain uncontrolled. For this group, deep brain stimulation (DBS) may be helpful.

The rationale for using deep brain stimulation (DBS) to treat epilepsy is that DBS disrupts regulatory feedback loops in the brain that allow seizures to develop and spread. By influencing these regulatory areas in the brain, electrical stimulation has the capacity to reduce or eliminate seizures that originate in portions of the brain that cannot safely be surgically removed. Vagus nerve stimulation (VNS) works in a similar way against seizures, but VNS disrupts the regulatory loops indirectly, while DBS disrupts the regulatory loops directly.

The thalamus is an appealing target for DBS to treat epilepsy because it has widespread connections to, and influences on, the cerebral cortex, which is the outer layer of the brain where seizures originate. Fourteen patients with various types of refractory epilepsy have been treated with stimulation of the anterior nucleus (AN) of the thalamus during the past several years. During the first 3 months of AN stimulation, the median seizure frequency reduction, relative to baseline, was 64%. Eight of the 14 patients (57%) had a 50% or greater decrease in seizure frequency (responders). Nine of the 14 patients had seizures presumed to arise from the temporal or frontal lobes. During the first 3 months, these 9 patients had a median 80% reduction in seizure frequency and 78% of them were responders. The AN was selected for stimulation because of its many connections to the "limbic system", a cortical system which is often a source of seizures.

Prior studies of thalamic stimulation for epilepsy (centromedian nucleus [CM]) The majority of the research addressing stimulation of the thalamic centromedian nucleus (CM) for the treatment of epilepsy has been reported by Velasco et al. (1-3). In 1987, the group published a paper in which 5 patients with generalized tonic-clonic seizures were implanted bilaterally. Stimulation was delivered 2 hours per day for 3 months. All patients experienced an 80-100% reduction in generalized tonic-clonic seizures and a 60-100% reduction in partial complex seizures. Much of the benefit observed continued beyond the 2-hour period of stimulation, suggesting that the stimulation resulted in a long-term change in thalamic activity.

In 1993, the same group published a report of 23 patients with externalized CM stimulators(2,3) (9 with generalized tonic-clonic seizures, 3 with focal motor and secondary generalized seizures, 5 with partial complex and secondary generalized seizures, and 6 with generalized tonic seizures and atypical absence seizures). These investigators found that stimulation resulted in a significant decrease in seizure frequency in the patients with tonic-clonic and partial motor seizures. However, no significant changes were observed in patients with complex partial seizures or generalized tonic seizures. Overall, 12 of the 23 patients had at least a 50% decrease in seizure frequency, and 1 patient was seizure free.

None of these studies from the Mexico City group (Velasco et al.) were blinded or controlled. However, in 1992, Fisher et al. (4) from John Hopkins reported a double-blind, controlled trial of CM stimulation. This treatment had no effects on the patients. Therefore, CM stimulation was abandoned and AN stimulation was undertaken instead.

Electroencephalograms (EEG) and thalamic stimulation for epilepsy An electroencephalogram (EEG) is a recording of brain wave electrical activity. The cerebral cortex nerve cells generate the EEG signal. The principal features of the EEG studied in patients with epilepsy are: 1) how rapidly and often the electrical signal changes amplitude ("frequency"), and 2) any abnormal excessive very brief unexpected electrical discharge ("spike-waves"). Spike-waves are the type discharges characteristic of patients with epilepsy.

Electrical stimulation of the CM nucleus of the thalamus has resulted in less EEG spike-waves (1-3). However, there have been no studies of EEG frequency in epilepsy patients receiving AN stimulation therapy.

For this study the investigators will record EEGs on computerized monitors. These recording machines are small portable computers (about the size of a "Walk-Man") which the patient wears for one hour. The brain-wave sensing electrodes are attached to the patients' scalp with a water-soluble temporary conducting glue. These monitors are placed on the patients in the EEG laboratory at New York Hospital-Cornell. The recorded EEG signal is downloaded to our EEG analysis computer. This is a routine test commonly performed to evaluate patients with epilepsy, and the ambulatory EEG in and of itself is not experimental in any way.

EEGs will be recorded at the following times relative to the DBS treatment for epilepsy: 1 month before stimulator implant, 1 month after stimulator implant (but before stimulator activation), after 3 months of DBS, after 6 months of DBS, and thereafter every 6 months or after stimulation setting changes.

The recorded EEGs will be mathematically analyzed, according to the following line of reasoning: Nerve cells in the thalamic AN connect to the cerebral cortex. AN activity (and AN stimulation) therefore may change how rapidly the electrical potentials of the cortex nerve cells change, which in turn may change the EEG frequency content. The investigators will utilize computer programs to determine the EEG frequency content, using a tool called "spectral analysis". The investigators will compare the spectral analysis between different time periods during the DBS treatment regimen.

Another feature the investigators will study is "EEG coherence". This is a computer-generated measure of how similar the brain wave frequencies are in different brain cortex regions. Since AN nerve cell activity regulates cortex nerve cell activity, AN stimulation may cause cortical activity in different regions of the brain to be more similar to each other. This type of change in cortical activity might be part of the mechanism of action of DBS against epilepsy. The investigators will compare the coherence analysis between different times during the DBS treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* To be scheduled to undergo deep brain stimulation therapy (DBS) in an attempt to treat intractable epilepsy

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
NA- observational study | 5 years appr.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Labar, MD, PhD, Principal Investigator — Weill Medical College at Cornell University
Locations (2):
- United States (2):
  - Weill Medical College at Cornell University - Comprehensive Epilepsy Center, New York, New York
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No